CLINICAL TRIAL: NCT06311851
Title: An Open-Label Pilot Study to Evaluate Efficacy and Safety of Bevacizumab Via Transarterial Chemoembolization (TACE) in Patients With Liver Metastases
Brief Title: Transarterial Chemoembolization (TACE) Plus Bevacizumab for Liver Metastases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pardis Noor Medical Imaging and Cancer Center (Other)
Responsible Party: Principal Investigator, Shahram Akhlaghpoor, Associate Professor of Vascular and Interventional Radiology, Pardis Noor Medical Imaging and Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNCC140201
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Metastatic Cancer; Liver Metastases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab Transarterial Chemoembolization (Experimental): The procedure commences with local disinfection and anesthesia, followed by a percutaneous right femoral artery puncture, performed using a modified Seldinger technique. A 5-F Simmons Ⅰ catheter was introduced through a vascular sheath and positioned in the common hepatic artery with the guidance of digital subtraction angiography to identify the tumor-supplying vessels. A 2.8-F microcatheter catheter was advanced into the vessel supplying the hepatic tumor. In cases of bilobar disease, the initial treatment focus was on the lobe with the greatest tumor burden, with the contralateral lobe addressed in a subsequent TACE session scheduled 4-6 weeks apart. In the standard TACE protocol ( hepaspheres are loaded with Irinotecan at 50 mg for colon metastases and Idarubicin at 10 mg for breast metastases), Bevacizumab 50 mg-loaded hepaspheres was added. The procedure was monitored under fluoroscopy until arterial flow stasis was achieved.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Infusion of Bevacizumab-loaded hepaspher through transarterial chemoembolization.

SUMMARY:
Trans arterial chemoembolization (TACE) has emerged as a treatment option for chemotherapy-refractory diseases in Liver metastases. By delivering chemotherapy agents directly to the tumor site, TACE can maximize local drug concentrations and reduce systemic adverse reactions. Bevacizumab is a monoclonal antibody that functions as an angiogenesis inhibitor. It works by slowing the growth of new blood vessels by inhibiting vascular endothelial growth factor A (VEGF-A). The application of Bevacizumab during TACE has not been reported. In this study, we will evaluate the the overall survival (OS)、efficacy, and safety of the application of Bevacizumab during TACE in patients with Liver Metastases by designing an open, single-arm phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of metastatic liver cancer via histological examination or a characteristic imaging profile on dynamic computed tomography (CT) scan or magnetic resonance imaging (MRI) without indications for surgical resection
* Eastern cooperative oncology group performance status (ECOGPS) of 0 or 1
* Liver function categorized as Child-Pugh class A or B
* Stable non-hepatic metastases, such as skeletal, pulmonary, or lymph node metastases
* Hepatic tumor burden below 70%
* Expected survival duration exceeding six months
* Laboratory findings meeting specific criteria, including platelet count >50×109 /L, hemoglobin >8.0 g/dL, ANC count ≥1.5 × 109/L, bilirubin <51 mmol/L, alanine and aspartate aminotransferase <3 times the upper limit of the normal range, and serum creatinine <1.5 times the upper limit of the normal range.

Exclusion Criteria:

* Active infection
* Presence of severe comorbidities, such as hepatic encephalopathy, refractory ascites, and esophageal variceal bleeding
* Prior liver resection
* Previous TACE therapy received at other healthcare facilities
* Poor performance status (ECOGPS > 1)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate | 6 months
  Percentage of patients who survived 6 months after inclusion
Objective response rate | 6 months
  The percentage of patients who achieved a complete or partial response at some point in their life

SECONDARY OUTCOMES:
Adverse event | 6 months
  Adverse event will be defined as the rate of patients who developed adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Pardis Noor Medical Imaging and Cancer Center, Tehran, Tehran Province, Iran